CLINICAL TRIAL: NCT04965246
Title: Trial Assessing Light Intensity Exercise on the Health of Older Breast Cancer Survivors
Acronym: TALIEHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Professor, Penn State Health Milton S Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PSCI 21-045
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Inflammation; Cognitive Impairment; Anxiety; Alcohol Drinking
MeSH Terms: conditions — Inflammation; Cognitive Dysfunction; Anxiety Disorders; Alcohol Drinking | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical activity (Experimental): the physical activity intervention will be structured to increase light-intensity aerobic physical activity, to achieve a total of 150 minutes per week. The intervention will also include weekly support calls from research staff to improve compliance to physical activity
  Interventions: Behavioral: Physical Activity
- Usual care (Other): Participants randomized to the usual care control group will serve as the control group for 15 weeks, and receive no intervention during this time.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Physical Activity — The physical activity program will focus on increasing physical activity, starting with a target of 100 minutes per week. The session durations will build over time to 150 minutes per week. Participants will be instructed to walk, or engage in other forms of light-intensity physical activity to achieve these goals. Participants will be instructed on the use of the ratings of perceived exertion scale (6-20). As the participants' health and fitness status improves, frequency, intensity, and session duration will be modified accordingly during weekly support calls. As participants will enter the study engaging in varying levels of physical activity, goals will be responsive to the most recent week's achieved minutes.
  Arms: Physical activity
Other: Usual Care — Participants in the usual care group will receive no intervention
  Arms: Usual care

SUMMARY:
The Trial Assessing Light-Intensity Exercise on the Health of Older Breast Cancer Survivors pilot randomized controlled trial aims to evaluate the efficacy of a home-based, light-intensity physical activity intervention among 56 obese, older adult breast cancer survivors, in comparison to a usual care control condition.

DETAILED DESCRIPTION:
The investigators will recruit 56 obese, older adult breast cancer survivors at least 1 year, and up to 10 years post-breast cancer treatment, and randomize them to either a 15 week light-intensity physical activity intervention, or usual care group.

Intervention: The participants will receive weekly support calls, and instructed to increase their light-intensity physical activity, to achieve at least 150 minutes per week. The frequency, intensity, time, and type of physical activity will be modified to maximize adherence and compliance. The support calls developed for this trial target older adults' capabilities, opportunities, and motivations for physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age 65-84 years
3. 1-10 years post-breast cancer treatment
4. Body mass index ≥30
5. ≥1 drink per week over the last month
6. ≥21 on the Telephone Interview For Cognitive Status
7. ≤7 on the Alcohol Use Disorder Identification Test
8. Fluent in written and spoken English
9. Must be able to provide and understand informed consent
10. Primary physician approval

Exclusion Criteria:

1. Body mass index <30
2. < 21 on the Telephone Interview for Cognitive Status
3. >7 on the Alcohol Use Disorder Inventory Test
4. Other neurological or major psychiatric disorders
5. Significant heart or lung disease
6. Limited life expectancy
7. Other factors that could potentially limit ability to participate fully in the intervention
8. Self-reporting achieving over 150 minutes of moderate-to-vigorous physical activity per week.

Ages: 65 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Markers of inflammation: C-reactive protein | Baseline
  A cytokine multiplex will assess markers of inflammation, including C-reactive protein
Markers of inflammation: C-reactive protein | 15 weeks
  A cytokine multiplex will assess markers of inflammation, including C-reactive protein

SECONDARY OUTCOMES:
Markers of inflammation-Interleukin 6 | Baseline
  A cytokine multiplex will assess markers of inflammation, including Interleukin 6
Markers of inflammation-Interleukin 6 | 15 weeks
  A cytokine multiplex will assess markers of inflammation, including Interleukin 6
Markers of inflammation-Tumor Necrosis Factor Alpha | Baseline
  A cytokine multiplex will assess markers of inflammation, including Tumor Necrosis Factor Alpha
Markers of inflammation-Tumor Necrosis Factor Alpha | 15 weeks
  A cytokine multiplex will assess markers of inflammation, including Tumor Necrosis Factor Alpha
The Functional Assessment of Cancer Therapy-Cognitive Function-Perceived Cognitive Impairments | Baseline
  The Functional Assessment of Cancer Therapy-Cognitive Function-Perceived Cognitive Impairments scores range from 0-72, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-Perceived Cognitive Impairments | 15 weeks
  The Functional Assessment of Cancer Therapy-Cognitive Function-Perceived Cognitive Impairments scores range from 0-72, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-Impact of perceived cognitive impairments on quality of life | Baseline
  The Functional Assessment of Cancer Therapy-Cognitive Function-Impact of perceived cognitive impairments on quality of life scores range from 0-16, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-Impact of perceived cognitive impairments on quality of life | 15 weeks
  The Functional Assessment of Cancer Therapy-Cognitive Function-Impact of perceived cognitive impairments on quality of life scores range from 0-16, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-comments from others | Baseline
  The Functional Assessment of Cancer Therapy-Cognitive Function-comments from others scores range from 0-16, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-comments from others | 15 weeks
  The Functional Assessment of Cancer Therapy-Cognitive Function-comments from others scores range from 0-16, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-perceived cognitive abilities | Baseline
  The Functional Assessment of Cancer Therapy-Cognitive Function-perceived cognitive abilities scores range from 0-28, higher scores indicate better quality of life.
The Functional Assessment of Cancer Therapy-Cognitive Function-perceived cognitive abilities | 15 weeks
  The Functional Assessment of Cancer Therapy-Cognitive Function-perceived cognitive abilities scores range from 0-28, higher scores indicate better quality of life.
Anxiety Symptoms-State-Trait Anxiety Inventory | Baseline
  State and trait anxiety are measured using the State and Trait subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol).The State-Trait Anxiety Inventory has 40 items, 20 items allocated to each of the subscales. State-Trait Anxiety Inventory varies from a minimum score of 20 to a maximum score of 80, higher scores indicate higher anxiety.
Anxiety Symptoms-State-Trait Anxiety Inventory | 15 weeks
  State and trait anxiety are measured using the State and Trait subscales of the State-Trait Anxiety Inventory (Spielberger, 2010, Corsini Encycl of Psychol).The State-Trait Anxiety Inventory has 40 items, 20 items allocated to each of the subscales. State-Trait Anxiety Inventory varies from a minimum score of 20 to a maximum score of 80, higher scores indicate higher anxiety.
Anxiety Symptoms-The Patient-Reported Outcomes Measurement Information System | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Anxiety subscale measures patient reported anxiety symptoms. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher anxiety
Anxiety Symptoms-The Patient-Reported Outcomes Measurement Information System | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Anxiety subscale measures patient reported anxiety symptoms. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher anxiety
Depressive Symptoms | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - depression subscale measures patient reported depressive symptoms. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher depression
Depressive Symptoms | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - depression subscale measures patient reported depressive symptoms. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher depression
Physical Function-The Patient-Reported Outcomes Measurement Information System | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - physical function subscale measures patient reported physical function. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher physical function
Physical Function-The Patient-Reported Outcomes Measurement Information System | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - physical function subscale measures patient reported physical function. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher physical function
Fatigue | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - fatigue subscale measures patient reported fatigue. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher fatigue.
Fatigue | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - fatigue subscale measures patient reported fatigue. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher fatigue.
Sleep Disturbance | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Sleep Disturbance subscale measures patient reported Sleep Disturbance. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviationof 10. Higher scores indicate higher Sleep Disturbance.
Sleep Disturbance-PROMIS-57 | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Sleep Disturbance subscale measures patient reported Sleep Disturbance. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Sleep Disturbance.
Ability to Participate in Social Roles and Activities | baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Ability to Participate in Social Roles and Activities subscale measures patient reported Ability to Participate in Social Roles and Activities. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Ability to Participate in Social Roles and Activities
Ability to Participate in Social Roles and Activities | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Ability to Participate in Social Roles and Activities subscale measures patient reported Ability to Participate in Social Roles and Activities. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Ability to Participate in Social Roles and Activities
Pain interference | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Pain interference subscale measures patient reported pain interference. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Pain interference
Pain interference | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Pain interference subscale measures patient reported pain interference. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Pain interference
Pain intensity | Baseline
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Pain interference subscale measures patient reported pain interference. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Pain intensity
Pain intensity | 15 weeks
  The Patient-Reported Outcomes Measurement Information System PROMIS®-57 Profile v2.1 - Pain interference subscale measures patient reported pain interference. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation of 10. Higher scores indicate higher Pain intensity
Alcohol consumption | Baseline
  A questionnaire probing the number of alcohol drinks consumed in the past 7 days
Alcohol consumption | 15 weeks
  A questionnaire probing the number of alcohol drinks consumed in the past 7 days
Physical Function-walk test | Baseline
  The six minute walking test will be administered to assess physical function. Participants will aim to walk as far as possible for 6 minutes.
  Further distances indicate greater physical function
Physical Function-walk test | 15 weeks
  The six minute walking test will be administered to assess physical function. Participants will aim to walk as far as possible for 6 minutes.
  Further distances indicate greater physical function
Mobile Monitoring of Cognitive Change | Week 1-2
  Ecological momentary assessment procedures for measuring both self-report and objective cognitive function will be used in 14 day bursts. These ecological momentary assessments protocols assess many of the same domains captured in other self-report and objective cognitive function measures, shortened and adapted for daily assessments.
Mobile Monitoring of Cognitive Change | Week 7-8
  Ecological momentary assessment procedures for measuring both self-report and objective cognitive function will be used in 14 day bursts. These ecological momentary assessments protocols assess many of the same domains captured in other self-report and objective cognitive function measures, shortened and adapted for daily assessments.
Mobile Monitoring of Cognitive Change | Week 14-15
  Ecological momentary assessment procedures for measuring both self-report and objective cognitive function will be used in 14 day bursts. These ecological momentary assessments protocols assess many of the same domains captured in other self-report and objective cognitive function measures, shortened and adapted for daily assessments.
Alcohol consumption-daily | Week 1-2
  Ecological momentary assessment procedures for measuring the number of drinks consumed in the past 24 hours will be assessed in 14 day bursts
Alcohol consumption-daily | Week 7-8
  Ecological momentary assessment procedures for measuring the number of drinks consumed in the past 24 hours will be assessed in 14 day bursts
Alcohol consumption-daily | Week 14-15
  Ecological momentary assessment procedures for measuring the number of drinks consumed in the past 24 hours will be assessed in 14 day bursts
Alcohol Use Disorder | Baseline
  The Alcohol Use Disorders Identification Test is a simple and effective method of screening for unhealthy alcohol use, defined as risky or hazardous consumption or any alcohol use disorder. A score of 8 or more is associated with harmful or hazardous drinking, a score of 13 or more in women, and 15 or more in men, is likely to indicate alcohol dependence.
Telephone Interview for Cognitive Status | Baseline
  The Telephone Interview for Cognitive Status is a brief, standardized test of cognitive functioning that was developed for use in situations where in-person cognitive screening is impractical or inefficient. The Telephone Interview for Cognitive Status will be used to screen for moderate-to-severe cognitive impairment. Scores 20 of lower indicate moderate-to-severe cognitive impairment
Demographics | Baseline
  Age, height, weight, family income, education level, age at diagnosis, time since diagnosis, injury history, diabetic status, and whether they are currently receiving treatment for mental health will be assessed at baseline
Acceptability-the proportion of older adults who agree to participate | Baseline
  The proportion of older adults who agree to participate among those deemed eligible.
Feasibility-the proportion of older adults who complete at least 50% of the physical activity intervention | Week 15
  The percentage of those randomized to the physical activity intervention that complete at least 50% of the physical activity intervention. Participants will be instructed by a project manager during weekly support calls to accumulate a specific amount of physical activity each week. Participants who self-report completing at least 50% of the physical activity, determined by the physical activity log, will be deemed compliant.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No